CLINICAL TRIAL: NCT05680454
Title: A Phase I Trial in Healthy Chinese Women Ages 18-45 to Evaluate the Safety and Tolerability Profile of Recombinant Nonavalent (Types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia Coli)
Brief Title: A Phase I Trial Evaluate the Safety and Tolerability Profile of HPV Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Health Guard Biotechnology, Inc (Industry)
Collaborators: Jiangsu Province Centers for Disease Control and Prevention (Network); National Institutes for Food and Drug Control, China (Other); Nanjing Sangruisi Pharmaceutical Technology Co., Ltd (Unknown); School of Public Health of Southeastern University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KLWS-V502-01
Record Dates: First submitted 2022-12-12; First posted 2023-01-11 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2022-12

CONDITIONS: Human Papillomavirus Infection
Keywords: CIN; VIN; VaIN; AIN; Cervical cancer; Vaginal cancer; vulvar cancer; Anal cancer; Genital warts
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Anus Neoplasms; Condylomata Acuminata | interventions — Papillomavirus Vaccines; Vaccines

STUDY DESIGN:
Intervention Model Description: The trial will be conducted in two stages:
  Stage 1: An open-label trial will be carried out in 40 healthy women ages 27-45 in the enrolment order of mid-dosage group followed by high-dosage group. Each group of 20 subjects will be administered the mid-, and high-dosage form respectively.
  Stage 2: A randomized and blinded (as to intra-dosage group) trial, with Gardasil9 as the positive control will be carried out in 120 healthy women ages 18-26 in the enrolment order of low-, mid-, and high-dosage groups. Each group of 40 subjects will be enrolled and randomized at a 3: 1 ratio to receive the investigational vaccine or positive control, respectively.
Who Masked: Participant, Investigator
Masking Description: The Sponsor, investigators and biostatisticians will remain blinded to subject allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Group of Investigational Vaccine (Experimental): For Low-dosage group, 0.5-mL suspension for injection, each 0.5-mL prefilled syringe dose contains L1 proteins of HPV types 6/11/16/18/31/33/45/52/58 in the amounts of 20μg、40μg、40μg、20μg、20μg、20μg、20μg、20μg, and 20μg respectively, totaling 220μg of antigens.
  For High-dosage group, 0.5-mL suspension for injection, each 0.5-mL prefilled syringe dose contains L1 proteins of HPV types 6/11/16/18/31/33/45/52/58 in the amounts of 30μg、40μg、80μg、60μg、30μg、30μg、30μg、30μg and 30μg respectively, totaling 360μg of antigens.
  For Mid-dosage group, 0.5-mL suspension for injection, each 0.5-mL prefilled syringe dose contains L1 proteins of HPV types 6/11/16/18/31/33/45/52/58 in the amounts of 30μg、40μg、60μg、40μg、20μg、20μg、20μg、20μg and 20μg respectively, totaling 270μg of antigens.
  Interventions: Biological: Recombinant Nonavalent (Types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia Coli)
- The Group of Active Control Vaccine (Active Comparator): Each 0.5-mL single-dose vial of GARDASIL9 contains approximately 30 mcg of HPV Type 6 L1 protein, 40 mcg of HPV Type 11 L1 protein, 60 mcg of HPV Type 16 L1 protein, 40 mcg of HPV Type 18 L1 protein, 20 mcg of HPV Type 31 L1 protein, 20 mcg of HPV Type 33 L1 protein, 20 mcg of HPV Type 45 L1 protein, 20 mcg of HPV Type 52 L1 protein, and 20 mcg of HPV Type 58 L1 protein, totaling 270 mcg of antigens.
  Interventions: Biological: Recombinant nonavalent Human Papillomavirus (Types 6,11,16,18,31,33,45,52,58) Vaccine

INTERVENTIONS:
Biological: Recombinant Nonavalent (Types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia Coli) — For Low-dosage group, a 3-dose regimen administered at months 0, 2 and 6. For Mid-dosage group, a 3-dose regimen administered at months 0, 2 and 6. For High-dosage group, a 3-dose regimen administered at months 0, 2 and 6.
  Arms: The Group of Investigational Vaccine
Biological: Recombinant nonavalent Human Papillomavirus (Types 6,11,16,18,31,33,45,52,58) Vaccine — A 3-dose regimen administered at months 0, 2 and 6.
  Arms: The Group of Active Control Vaccine

SUMMARY:
This study is to evaluate the safety and tolerability profile of Recombinant Nonavalent (Types 6/11/16/18/31/33/45/52/58) Human Papillomavirus (HPV) Vaccine (Escherichia Coli) in healthy women ages 18-45

DETAILED DESCRIPTION:
This is a single-centre, dose-escalating, randomized, blinded and active controlled trial in healthy Chinese women ages 18-45. The positive control is Recombinant nonavalent Human Papillomavirus (Types 6,11,16,18,31,33,45,52,58) Vaccine.

The trial will be conducted in two stages:

Stage 1: A single-center, open-label trial will be carried out in 40 healthy women ages 27-45 in the enrolment order of mid-dosage group followed by high-dosage group. Each group of 20 subjects will be administered the mid-, and high-dosage form, respectively, to preliminarily evaluate the safety profile of the investigational vaccine.

First, the 20 subjects in the mid-dosage group will be sequentially enrolled as two batches of 5 and 15 subjects, respectively, at an enrolment interval of no less than 3 days. One week after vaccinating all the 20 subjects in the mid-dosage group, upon confirmation of the safety profile of the investigational vaccine as acceptable, 20 subjects for the higher dosage-group will be enrolled subsequently in the same manner as those in the mid-dosage group.

Subjects in each dosage group will receive a 3-dose regimen at months 0, 2 and 6. Safety of the investigational vaccine will be assessed for 30 days following each injection, and SAE will be reported for the duration of the study. In total there will be 12 scheduled visits for subjects in each dosage group throughout the study.

One week after vaccinating all the 40 subjects in stage 1, if the safety profile of the investigational vaccine is confirmed to be acceptable, the study may proceed to stage 2.

Stage 2:

A phase I, single-center, dose-escalating, randomized and blinded (as to intra-dosage group) trial, with Gardasil9 as the positive control will be carried out in 120 healthy women ages 18-26 in the enrolment order of low-, mid-, and high-dosage groups. Each group of 40 subjects will be enrolled and randomized at a 3: 1 ratio to receive the investigational vaccine or positive control, respectively (that is, 10 of the subjects in each dosage group will receive the positive control).

Firstly, the 40 subjects in the low-dosage group will be sequentially enrolled as four batches of 5, 10, 10 and 15 subjects, respectively, at an enrolment interval of no less than 3 days to get the first dose of the low-dosage investigational vaccine or positive control. Then, one week after vaccinating all the 40 subjects in the low-dosage group, upon confirmation of the safety profile of the investigational vaccine as acceptable, 40 subjects will be enrolled subsequently into the mid-dosage group in the same manner as those in the low-dosage group. Again, one week after vaccinating the 40 subjects in the mid-dosage group, if the safety profile of the investigational vaccine continues to be acceptable, another group of 40 subjects receiving the high-dosage investigational vaccine or positive control will be enrolled subsequently in the same manner as those in the low-dosage group.

In both stage 1 and stage 2 of the phase I study, 5 ml of non-anticoagulative blood will be collected from trial subjects prior to dose 1 and at Month 3 and Month 7 post dose 1 to determine the levels of neutralizing antibodies and IgG antibodies to the vaccine HPV types.

ELIGIBILITY:
Inclusion Criteria:

Stage 1:

1. Female subjects 27-45 years of age (inclusive of 27 and 45 years of age);
2. Subjects decided to be healthy by the principal investigator in accordance with such trial subjects' medical history and physical examination results;
3. Subjects who understand and agree to comply with the study procedures and provide written informed consent;
4. Subjects who are able to comply with protocol-specified requirements;
5. Subjects with negative urine pregnancy test result at screening;
6. Subjects with no childbearing potential (e.g. females who have undergone bilateral tubal ligation, hysterectomy, bilateral oophorectomy, etc.), or subjects with childbearing potential who have agreed to abstain from any sexual activity that could result in pregnancy or practice adequate contraception for at least 28 days prior to the first dose and throughout the study;
7. Subjects with axillary temperature≤37.0℃.

Stage 2:

1. Female subjects 18-26 years of age (inclusive of 18 and 26 years of age);
2. Subjects decided to be healthy by the principal investigator in accordance with such trial subjects' medical history and physical examination results;
3. Subjects who understand and agree to comply with the study procedures and provide written informed consent;
4. Subjects who are able to comply with protocol-specified requirements;
5. Subjects with negative urine pregnancy test result at screening;
6. Subjects with no childbearing potential (e.g. females who have undergone bilateral tubal ligation, hysterectomy, bilateral oophorectomy, etc), or subjects with childbearing potential who have agreed to abstain from any sexual activity that could result in pregnancy or practice adequate contraception for at least 28 days prior to the first dose and throughout the study;
7. Subjects with axillary temperature≤37.0℃.

Exclusion Criteria:

The same exclusion criteria apply to both stage 1 and stage 2

1. Women who are pregnant or breastfeeding, or planning for pregnancy in the following 7 months;
2. Women who have received other HPV vaccine(s) prior to dose 1 of the interventions;
3. Women who have received an investigational or unregistered drug or vaccine within 28 days prior to the first dose of the interventions, or plan to receive an investigational or unregistered drug or vaccine during the study;
4. Women who have known allergy history or who are allergic to any component of the interventions, such as penicillin and amikacin;
5. Women with a history of severe adverse reactions to previous vaccinations, such as allergies, urticaria, dyspnea, angioneurotic edema, or abdominal pain;
6. Women who have an autoimmune disease or immunodeficiency, are HIV positive, or have primary diseases in vital organs;
7. Women who have asthma that is unstable and requires urgent care, hospitalization and the use of oral or intravenous corticosteroids during the past two years;
8. Women who have diabetes mellitus (type I or II), with the exception of gestational diabetes;
9. Women with a history of thyroidectomy or thyroid diseases that required medical care within the past 12 months.;
10. Women with serious angioedema episodes within the past 3 years or requiring medical care over the past 2 years;
11. Women who have hypertension over 145/95 mm Hg at enrolment despite being treated by medication;
12. Women with coagulation disorders as diagnosed by a doctor (e.g. coagulation factor deficiency, coagulopathy, or platelet disorder) or coagulation difficulty;
13. Women with active malignancy, or treated malignancy for which there is no reasonable assurance of sustained cure, or malignancy that is likely to recur during the study;
14. Women with a history of epilepsy other than epilepsy with febrile seizures under two years of age, epilepsy secondary to alcohol use 3 years prior to alcohol withdrawal, or a singular epileptic seizure not requiring treatment within the past 3 years;
15. Women with the condition of asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen;
16. Women with a history of systematic chemotherapy in the past 5 years, a history of immunosuppressive therapy and cytotoxic therapy, and treatment with inhaled corticosteroids within the past 6 months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis), and women who received blood products in the 3 months prior to vaccination with the interventions;
17. Women who received a live attenuated vaccine during the 28 days prior to vaccination with the interventions; Women who received a subunit or inactivated vaccine, such as pneumococcal vaccine, or underwent antianaphylactic treatment during the 14 days prior to vaccination with the interventions;
18. Women who received a subunit or inactivated vaccine, such as pneumococcal vaccine, or underwent antianaphylactic treatment during the 14 days prior to vaccination with the interventions;
19. Women who are currently on an anti-TB prophylaxis or therapy;
20. Women who had fever (with axillary temperature≥38.0℃) during the 3 days prior to vaccination with the interventions or onset of any acute illness that required the use of antibiotics and antiviral treatment within the past 5 days;
21. Women with psychiatric conditions that preclude compliance with the protocol, or women with past or present psychoses, past or present bipolar disorder that has not been well controlled over the past 2 years, or women who are on medication for psychoses, or women who had suicidal thoughts/tendency in the past 5 years prior to enrolment;
22. Women with any medical, psychological or social conditions, or for occupational reasons or otherwise as judged by the principal investigator, that preclude participation in the study, or compromise a subject's ability to give informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Percentage of adverse reaction(s) within 7 days post any dose of the interventions. | 0-7 months
  Percentage of subjects with 1 or more injection-site or non-injection-site (systemic) adverse reaction(s) within 7 days post any dose of the interventions.

SECONDARY OUTCOMES:
Percentage of adverse event(s) within 30 days post any dose of the interventions | The 3rd day after each injection
  Percentage of subjects with 1 or more injection-site or non-injection-site (systemic) adverse event(s) within 30 days post any dose of the interventions
Percentage of abnormal blood routine indexes, coagulation time and blood biochemical indexes | The 3rd and 7th month after immunization
  Percentage of subjects with abnormal blood routine indexes (concentrations of hemoglobin, white blood cells count), abnormal coagulation time (PT, APTT), and abnormal blood biochemical indexes (creatinine, alanine aminotransferase, aspartate aminotransferase) 3 days after any any dose of the interventions.
Percentage of serious adverse event(s) | 0-7 months
  Percentage of subjects with serious adverse event(s) for the duration of the study (about 7 months).
Levels of neutralization antibodies against each vaccine HPV type (6/11/16/18/31/33/45/52/58) | The 7th month after immunization
  Levels of neutralization antibodies against each vaccine HPV type (6/11/16/18/31/33/45/52/58) one month post dose 3 (Month 7) among trial subjects.
Percentage of subjects positive for neutralization antibodies against each vaccine HPV type (6/11/16/18/31/33/45/52/58) | The 7th month after immunization
  Percentage of subjects positive for neutralization antibodies against each vaccine HPV type (6/11/16/18/31/33/45/52/58) one month post dose 3 (Month 7) among trial subjects.
Levels of IgG antibodies | The 7th month after immunization
  Levels of IgG antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) one month post dose 3 (Month 7) among trial subjects.
Seropositive rates of IgG antibodies | The 7th month after immunization
  Seropositive rates of IgG antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) one month post dose 3 (Month 7) among trial subjects.
Levels of neutralizing antibodies | The 3rd month after immunization
  Levels of neutralizing antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at month 3 post dose 1 among trial subjects.
Levels of IgG antibodies | The 3rd month after immunization
  Levels of IgG antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at month 3 post dose 1 among trial subjects.
Seropositive rates of neutralizing antibodies | The 3rd month after immunization
  Seropositive rates of neutralizing antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at month 3 post dose 1 among trial subjects.
Seropositive rates of IgG antibodies | The 3rd month after immunization
  Seropositive rates of IgG antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at month 3 post dose 1 among trial subjects.
Seroconversion rates of neutralizing antibodies | The 3rd and 7th month after immunization
  Seroconversion rates of neutralizing antibodies Seroconversion rates of neutralizing antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at Month 3 and Month 7 post dose 1, respectively, among trial subjects.
Seroconversion rates of IgG antibodies | The 3rd and 7th month after immunization
  Seroconversion rates of IgG antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at Month 3 and Month 7 post dose 1, respectively, among trial subjects.
Fold increases in levels of neutralizing antibodies and IgG antibodies | The 3rd and 7th month after immunization
  Fold increases in levels of neutralizing antibodies and IgG antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at Month 3 and Month 7 post dose 1, respectively, among trial subjects.
Levels of neutralizing antibodies | Before immunization, and the 3rd and 7th month after immunization
  Levels of neutralizing antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at Month 3 and Month 7 post dose 1, respectively, among trial subjects who were negative for antibodies to the corresponding HPV type (HPV 6/11/16/18/31/33/45/52/58) prior to dose 1
Levels of IgG antibodies | Before immunization, and the 3rd and 7th month after immunization
  Levels of IgG antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at Month 3 and Month 7 post dose 1, respectively, among trial subjects who were negative for antibodies to the corresponding HPV type (HPV 6/11/16/18/31/33/45/52/58) prior to dose 1
Seroconversion rates of neutralizing antibodies | Before immunization, and the 3rd and 7th month after immunization
  Seroconversion rates of neutralizing antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at Month 3 and Month 7 post dose 1, respectively, among trial subjects who were negative for antibodies to the corresponding HPV type (HPV 6/11/16/18/31/33/45/52/58) prior to dose 1
Seroconversion rates of IgG antibodies | Before immunization, and the 3rd and 7th month after immunization
  Seroconversion rates of IgG antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at Month 3 and Month 7 post dose 1, respectively, among trial subjects who were negative for antibodies to the corresponding HPV type (HPV 6/11/16/18/31/33/45/52/58) prior to dose 1
Fold increases in neutralizing antibodies | Before immunization, and the 3rd and 7th month after immunization
  Fold increases in neutralizing antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at Month 3 and Month 7 post dose 1, respectively, among trial subjects who were negative for antibodies to the corresponding HPV type (HPV 6/11/16/18/31/33/45/52/58) prior to dose 1
Fold increases in IgG antibodies | Before immunization, and the 3rd and 7th month after immunization
  Fold increases in IgG antibodies to each vaccine HPV type (6/11/16/18/31/33/45/52/58) at Month 3 and Month 7 post dose 1, respectively, among trial subjects who were negative for antibodies to the corresponding HPV type (HPV 6/11/16/18/31/33/45/52/58) prior to dose 1

CONTACTS AND LOCATIONS:
Overall Officials: Yongjiang Liu, Bachelor, Study Chair — Beijing Health Guard Biotechnology, Inc
Locations (1):
- CDC, Jiangsu Province, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
No informed consent was obtained to disclose the subject's data and sample test results.